CLINICAL TRIAL: NCT02827955
Title: Evaluation of Bilateral Gamma Knife Thalamotomy in Patients Presenting With Severe Essential Tremor
Acronym: VIMBIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-38; 2013-A01289-36 (Other: IDRCB); 2013-38 (Other: APHM)
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Patients With Parkinson's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bilateral thalamotomy radiosurgery (Experimental): Gamma Knife radiosurgery bilateral
  Interventions: Device: Gamma Knife® radiosurgery bilateral

INTERVENTIONS:
Device: Gamma Knife® radiosurgery bilateral

SUMMARY:
Essential tremor (ET) is the most frequent movement disorder. Its prevalence is about 1/200 implying that at least 300 000 peoples are concerned in France. Its frequency increase with age (14% of patients 65 yo). The diagnostic criteria are postural and kinetic tremor that can be associated with head/voice tremor. ET induces a social impairment but also difficulties to perform any task requiring dexterity. With time, tremor can be so severe that every activity of daily living is impaired with loss of autonomy.

Treatment such as betablockers, primidone or antiepileptics might have some efficacy at the beginning. But as the severity of the tremor increases, there is lack of efficacy. Deep Brain stimulation (DBS) of the ventral intermediate nucleus (VIM) of the thalamus can be proposed. However, in case of medical or surgical contra-indication, Gamma Knife (GK) radiosurgery thalamotomy can be an alternative option.

Patients will be included with a minimum of 12 months after having the first thalamotomy (Gamma Knife 1) (done on the most annoying side) subject to no significant deterioration in cognitive assessment, voice assessment and balance and postural assessment or neuroradiological abnormality.

Patients will be assessed with Magnetic resonance imaging (MRI) cerebral, clinical assessment (tremor rating scale) impairment of activity of daily living, neuropsychological evaluation, voice assessment and balance and postural assessment.

The second thalamotomy (Gamma Knife 2) will be proposed and a monitoring at M6 and M12 will be done.

This study will demonstrate the feasibility and tolerance of bilateral GK radiosurgery thalamotomy in ET patients with severe impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential tremor defined criteria Consensus statement of the movement Disorder Society on Classical Essential Tremor (1998), with trembling of the upper limbs causing functional impairment justifying surgical therapy.
* Man or woman aged 20 to 85 years.
* Patient having an absolute contraindication against or on Deep Brain Stimulation (DBS) of the VIM.
* Patient who received a first effective unilateral thalamotomy on tremor with a satisfactory clinical outcome (no cognitive impairment, lack of postural disorder Musculoskeletal severe lack of dysarthria). The first effective thalamotomy will be characterized by an improved score of tremor ≥ 45% and improved functional gene ≥ 50%.
* Patient who received a first unilateral thalamotomy with satisfactory radiological evolution. Unsatisfactory radiological evolution will be characterized by a contrast uptake> 350 mm3 one year with edema on T2 and Flair sequences extended beyond the internal capsule.
* Patient requiring contralateral treatment because of the severity of the tremor and functional impairment.
* Patient affiliated to a social protection scheme.
* Patient who understood and signed the informed consent form (signature of a third person possible when the patient is unable to read and / or write but in a state to give consent).

Exclusion Criteria:

* Patient with against-indication for performing a brain MRI (pacemaker, intracranial metallic objects etc.)
* Patient with an against-indication to radiosurgical treatment (prior treatment with cerebral radiotherapy)
* Pregnant or lactating women
* Women of childbearing potential unless

  1. surgical sterilization
  2. use of effective contraception (intrauterine device or method more hormonal barrier method), and requiring to present a test pregnancy by assaying the negative serum with chorionic gonadotrope hormon (CGH) when selecting and accept to remain under the current form of contraception for the duration of the study (in women past menopause should be amenorrheic for at least 12 months to be considered as no longer able to bear a child).
* simultaneous participation in another clinical trial or exclusion period of a previous clinical trial.
* vulnerable persons: minors, protected adults (guardianship) and Major unable to consent.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
evaluation of cognitive tolerance | 36 months
  Define therapeutic technique "acceptable" in cognitive tolerance level by the Mini Mental State scale (MMS), 10% of subjects decrease their MMS over 2 points.

CONTACTS AND LOCATIONS:
Overall Officials: Jean REGIS, PUPH, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No